CLINICAL TRIAL: NCT03203993
Title: China Local BRCA Testing and Exploration of Ovarian Cancer Treatment Outcomes of Different BRCA Status in Newly Diagnosed Epithelial Ovarian Cancer Patients
Brief Title: China Ovarian Cancer BRCA Testing Study
Acronym: CRONUS
Status: Terminated | Type: Observational
Why Stopped: Failure to obtain HGR approval.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133FR00117
Record Dates: First submitted 2017-06-23; First posted 2017-06-29 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Ovarian Cancer
Keywords: BRCA mutation
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, multi-center, observational study, the primary objective is to evaluate the prevalence of gBRCA/sBRCAm in newly diagnosed ovarian cancer patients and explore ovarian cancer treatment outcomes of different BRCAm status

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational study that will enroll consecutive patients with a confirmed diagnosis of epithelial ovarian cancer, fallopian tube, or peritoneal cancer and who consent to a blood draw, a tissue sample analysis, and follow up for collection of data. 900 newly diagnosed ovarian cancer patients will be enrolled and evaluated for Breast Cancer Susceptibility genes BRCA1 and BRCA2 germline and somatic mutations (BRCAm). Approximately 170 BRCAm positive patients and 170 negative patients will be followed in the Follow-up Period. This study aims to answer very important questions regarding the prevalence of gBRCAm and sBRCAm in a population of newly diagnosed ovarian cancer patients, and the relationship of these mutations to patient treatment and clinical outcomes. These answers may be extremely helpful in the counseling and treatment of genetic risk in these populations and may aid in making treatment decisions in the future.

ELIGIBILITY:
Inclusion Criteria:

* Be able and willing to sign the informed consent form (ICF)
* Female aged 18 years or over
* Have histologically confirmed new diagnosis of Federation of Gynecology and Obstetrics (FIGO) stage III or IV ovarian epithelial, primary peritoneal, or fallopian tube cancer made by one or more of the following:

  * standard staging laparotomy including bilateral salpingo-oophorectomy, omentectomy, and lymph node sampling and debulkingand/or
  * surgical resection and radiographic evidence consistent with Stage III or IV ovarian cancer
  * biopsy with radiographic evidence consistent with Stage III or IV ovarian cancer
* Have availability of paraffin-embedded archivedtumor tissue block (preferred) or,if a block is not possible, a minimum of twenty 5-μm unstained sections. (Tumor tissue should be archived at diagnosis. 10 slides is utilized for sBRCA testing after the enrolment. Another 10 slides is utilized for exploratory evaluation of HRR gene mutations in a retrospective way.)
* Have a diagnosis that is within 60 days of informed consent

Exclusion Criteria:

* Have a diagnosis of additional concurrent malignancies or previous diagnosis of another malignancy with current evidence of residual disease
* Have a diagnosis of other severe acute or chronic medical or psychiatric conditions that may increase the risk associated with study participation or may interfere with the interpretation of the study results and, in the judgement of the Investigator, would make the patient inappropriate for enrollment in this study
* Be currently participating in any other clinical trial for first-line treatment of ovarian cancer
* Be a patient who, in the judgement of the Investigator, would be inappropriate for enrollment in this study

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: newly diagnosed epithelial ovarian cancer patients
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of newly diagnosed ovarian cancer patients with gBRCA and sBRCA mutations | 1 year
  To evaluate the prevalence of gBRCA mutation and sBRCA mutation in newly diagnosed ovarian cancer patients

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 18 months
  To describe ovarian cancer treatment outcomes in patients during the Follow up Period in terms of PFS
Overall survival (OS) | up to 5 years
  To describe ovarian cancer treatment outcomes in patients during the Follow up Period in terms of OS

OTHER OUTCOMES:
Proportion of newly diagnosed ovarian cancer patients with HRR gene mutations | 1 year
  To evaluate the prevalence of homologous recombination repair (HRR) gene mutations in newly diagnosed ovarian cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Jinghe Lang, Dr, Study Chair — Peking Union Medical College Hospital
Locations (13):
- China (12):
  - Research Site, Hefei, Anhui
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Chongqing, Chongqing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Zhengzhou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Jinan, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Hangzhou, Zhejiang
- Research Site, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca has a long-standing commitment to making information about our clinical research publicly available. We believe that transparency enhances the scientific understanding of how our medicines work and is in the medical interest of our patients.
  We publish information on the registration and results of all new and ongoing AstraZeneca sponsored clinical trials for all products in all phases, including marketed medicines, drugs in development and drugs whose further development has been discontinued. We post results, irrespective of whether they are favourable or unfavourable to AstraZeneca.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.